CLINICAL TRIAL: NCT05899309
Title: Precision Medicine to Predict the Trajectory of Liver Cirrhosis : Prospective Cohort Study
Brief Title: Precision Medicine to Predict the Trajectory of Liver Cirrhosis: Prospective Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Changi General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2021/2815
Record Dates: First submitted 2023-05-24; First posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Liver Cirrhosis; Metabolic Syndrome; Spleen; Fibrosis; Frailty
Keywords: liver cirrhosis; Metabolic syndrome; Cardiovascular events
MeSH Terms: conditions — Liver Cirrhosis; Metabolic Syndrome; Fibrosis; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — 6 mls of blood , 20 ml of urine and 1 gm of stool for research will be taken at Visit 1 and 3 . If there is decompensation 5 mls of blood will be obtain at each event.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Liver cirrhosis with metabolic syndrome: Liver cirrhosis patients with metabolic syndrome on standard treatment
  Interventions: Diagnostic Test: liver and spleen stiffness test and laboratory test
- Liver cirrhosis without metabolic syndrome: Liver cirrhosis patients without metabolic syndrome on standard treatment
  Interventions: Diagnostic Test: liver and spleen stiffness test and laboratory test

INTERVENTIONS:
Diagnostic Test: liver and spleen stiffness test and laboratory test — Diagnosis of cirrhosis can be based on liver biopsy,radiological ,clinical or liver stiffness measurement (LMS)

SUMMARY:
Preventing decompensation is a key endpoint in the management of compensate cirrhosis patients. The known factors that increases the risk of decompensation include the presence of clinically significant portal hypertension (CSPH) and the control of primary etiology of cirrhosis. Other factors which may influence the progression of cirrhosis included the presence of metabolic syndrome (diabetes mellitus and obesity), frailty, concomitant medications (statin, non-selective beta-blocker) were not well understood. Investigators aim to perform a pilot, observational study to study various baseline factors in relation to the clinical outcome of cirrhosis patients in a prospective follow up.

DETAILED DESCRIPTION:
All patient who fulfilled eligibility criteria will be consented and recruited. The study will last up to 3 years or up to 7 assessment and 7 visits All subjects will be followed every 6 monthly for study outcome from recruitment, biosamples (blood,urine and stool), elastography, quality of life questionnaire and frialty assessment were done at baseline. Completion of Sit to stand , handgrip and 6 minute walking test at baseline and Visit 3.All visits will be follow up on study outcome (liver-related events ,metabolic related outcome and cardiovascular related outcomes.). During decompensation (decrease in liver function ) .Collection of research leftover blood,urine and stool samples if applicable.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21 to 90 years with the diagnosis of liver cirrhosis (regardless of etiology)
* Consent to participate in the study

Exclusion Criteria:

* Terminal malignancy. Subjects with prognosis < 3 months.
* Patient refusal or unable to commit to study follow-up

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Personalize risk stratification in an unmet need because compensated cirrhosis patients has heterogeneous risk of deterioration.
  With growing prevalence of obesity, there are more and more cirrhosis patients having metabolic syndrome. The impart of metabolic syndrome among cirrhosis patients remain unclear.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-05-23 (Actual); Primary Completion 2023-12-12 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Liver related events | 3 years
  Determine the rate of liver related events with and without metabolic syndrome

SECONDARY OUTCOMES:
Progression of cirrhosis | 3 years
  To determine the proportion of patients with cirrhosis progression (stage as defined by D' Amico method).
Cardiovascular events | 3 years
  Determine the rate of cardiovascular events with and without metabolic syndrome
Baseline cirrhosis features | 3 years
  Baseline differences (clinical, immunological and metabolomic differences) and liver stiffness and spleen stiffness measured using vibration on controlled transient elastography (in kPa) between cirrhosis patients with and without metabolic syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Yu Jun Wong, MD, Principal Investigator — Changi General Hospital
Locations (1):
- Changi General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harris PS, Hansen RM, Gray ME, Massoud OI, McGuire BM, Shoreibah MG. Hepatocellular carcinoma surveillance: An evidence-based approach. World J Gastroenterol. 2019 Apr 7;25(13):1550-1559. doi: 10.3748/wjg.v25.i13.1550. PMID 30983815
- [Background] Chang PE, Wong GW, Li JW, Lui HF, Chow WC, Tan CK. Epidemiology and Clinical Evolution of Liver Cirrhosis in Singapore. Ann Acad Med Singap. 2015 Jun;44(6):218-25. PMID 26292950